CLINICAL TRIAL: NCT06812221
Title: A Phase 1/2 Randomized, Double-Blind, Placebo-Controlled Trial of Multiple Sublingual 5-MeO-DMT Microdoses for Reducing Anxiety and/or Depression in Patients With Mild Cognitive Impairment.
Brief Title: Efficacy of Sublingual 5-MeO-DMT for Reducing Anxiety and Depression in MCI
Acronym: 5-MeO-DMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomind Labs Inc. (Industry)
Collaborators: Hospital Descentralizado Dr. Marcial V. Quiroga (Unknown); Universidad Católica de Cuyo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMND08-03
Record Dates: First submitted 2024-12-10; First posted 2025-02-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Anxiety State; Depression Anxiety Disorder
Keywords: double blind placebo-controlled; Phase I/II clinical trial; ramdomized; sublingual administration; 5-MeO.DMT; anxiety; Depression; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Anxiety Disorders; Depression | interventions — Administration, Sublingual; Vital Signs

STUDY DESIGN:
Intervention Model Description: This Phase I/II clinical trial uses a randomized, double-blind, placebo-controlled design to evaluate the effects of 6 mg sublingual 5-MeO-DMT on individuals with Mild Cognitive Impairment (MCI). Participants will be randomly assigned to either the active treatment group or the placebo group, each consisting of 10 participants. The trial will last 4 weeks, with weekly doses administered under supervision. Primary outcomes include assessments of cognitive function (via ACE III and IFS) and mood (via BDI II and STAI). Safety will be closely monitored through regular checks on vital signs, ECGs, biochemical markers, and psychological evaluations. The goal is to assess the cognitive and psychological effects of 5-MeO-DMT, contributing to the understanding of its potential as a treatment for MCI-related symptoms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Arm 1: 6 mg 5-MeO-DMT Sublingual Administration (Experimental): In this arm, participants will receive a single sublingual dose of 6 mg of 5-MeO-DMT once a week for four consecutive weeks. This dosage aims to assess the potential therapeutic effects of 5-MeO-DMT in reducing anxiety and depression symptoms in individuals with Mild Cognitive Impairment (MCI). The 6 mg dose is selected to avoid inducing strong psychedelic effects, focusing on emotional well-being improvement. Participants will undergo standardized psychiatric assessments, such as STAI and BDI II, to measure changes in mood and anxiety levels. Additionally, neurocognitive assessments, including the Phonological Verbal Fluency Test (FAS), Paced Auditory Serial Addition Test (PASAT), and Digit Span Scale (DSS), will evaluate cognitive effects on executive function, processing speed, and working memory. Participants will be monitored closely for any adverse effects, changes in vital signs, and alterations in emotional or cognitive states throughout the study.
  Interventions: Drug: Sublingual administration; Procedure: Electroencephalography; Diagnostic Test: Biochemical mesurements; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: Vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments
- : Arm 2: Placebo Sublingual Administration (Experimental): Participants will receive a placebo formulation that mirrors the appearance, taste, and administration method of the 5-MeO-DMT doses but contains no active ingredient. This group will serve as the comparator, allowing the effects of the active 5-MeO-DMT treatment to be evaluated. Participants will undergo the same psychiatric and neurocognitive assessments as those in the experimental arm, including the STAI, BDI II, DASS-21, and cognitive tests. The placebo group will provide essential baseline data on mood, anxiety, and cognitive function, helping to determine whether observed changes in the experimental arms are due to the active drug. Monitoring for adverse events and changes in emotional or cognitive states will also be conducted in this group. The differences between this group and the 5-MeO-DMT arms will help establish the efficacy of 5-MeO-DMT for improving mood and cognitive function in individuals with MCI.
  Interventions: Drug: Sublingual administration; Procedure: Electroencephalography; Diagnostic Test: Biochemical mesurements; Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects; Diagnostic Test: Vital signs; Diagnostic Test: Cognitive Assessments; Diagnostic Test: Psychiatric Assessments

INTERVENTIONS:
Drug: Sublingual administration — Participants will receive a sublingual dose of 5-MeO-DMT or placebo, once a week for four consecutive weeks.
Procedure: Electroencephalography — Conducting baseline electroencephalography and during the consumption of the corresponding dose.
Diagnostic Test: Biochemical mesurements — Biochemical determinations will be performed to assess hematological, renal, hepatic, cardiac, and cellular lysis functions. The biochemical markers that will be measured include red blood cells, hematocrit, hemoglobin, glycated hemoglobin, white blood cells, microalbuminuria (urine albumin/creatinine ratio), and various serum markers such as cortisol, glucose, urea, serum creatinine, total cholesterol, HDL, LDL, triglycerides, AST, ALT, lactate dehydrogenase (LDH), creatine kinase (CK), CK-MB, and C-reactive protein.
Diagnostic Test: Acute Subjective Ratings of Psychedelic Effects — To determine the intensity of the acute effects experienced by subjects, retrospective ratings will be collected 1 hour after 5-MeO-DMT or placebo exposure. Subjective ratings will include the Peak Experience Scale (PES), the Ego Dissolution Inventory (EDI), and the Mystical Experiences Questionnaire (MEQ).
Diagnostic Test: Vital signs — Vital signs, including blood pressure, heart rate, oxygen saturation, respiration rate, body temperature, and electrocardiograms (ECGs), will be monitored over the six weeks of the treatment.
Diagnostic Test: Cognitive Assessments — Cognitive assessments will evaluate the effects of sublingual 5-MeO-DMT on cognitive functions. Participants will complete the Phonological Verbal Fluency Test (FAS) to assess executive function, the Paced Auditory Serial Addition Test (PASAT) to evaluate processing speed, and the Digit Span Scale (DSS) to measure attention span and working memory. These tests will be administered at baseline, during treatment, and post-treatment to monitor any cognitive changes in response to either a 6 mg dose of 5-MeO-DMT or placebo. This will help determine how the intervention may affect cognitive processing, memory, and attention.
Diagnostic Test: Psychiatric Assessments — Psychiatric evaluations will be conducted to assess the emotional and psychological effects of sublingual 5-MeO-DMT. Participants will complete the Beck Depression Inventory II (BDI II) to measure mood and depressive symptoms, the State-Trait Anxiety Inventory (STAI) to evaluate state anxiety, and the Depression, Anxiety, and Stress Scale (DASS-21) to assess stress levels. Additionally, the Suicidal Ideation Scale (SSI) will be used to monitor any changes in suicidal ideation throughout the study. These psychiatric assessments will be administered at multiple time points during the study to evaluate the potential therapeutic effects of 5-MeO-DMT in improving mood, anxiety, and overall psychological well-being.

SUMMARY:
This Phase I/II clinical trial aims to test the effectiveness of a new sublingual formulation of 5-MeO-DMT in reducing symptoms of anxiety, depression, and cognitive decline in individuals with mild to moderate Alzheimer's disease. The study will include participants who have a Clinical Dementia Rating (CDR) score between 0.5 and 1, indicating mild to moderate cognitive impairment, and who meet specific educational and cognitive criteria. Participants must have an ACE-III score of ≤86 for individuals with a high level of education (≥12 years) or <62 for those with a low educational level (≤12 years). Additionally, participants must show moderate to high levels of anxiety, as indicated by the State-Trait Anxiety Inventory (STAI), with STAI-S (State) scores ≥20 for men and ≥23 for women, and STAI-T (Trait) scores ≥20 for men and ≥26 for women. Participants also need to exhibit moderate to severe depressive symptoms, as indicated by a Beck Depression Inventory (BDI) score of ≥21.

To ensure that participants are cognitively functional but showing signs of impairment, they are assessed with the CDR and ADLQ scales to confirm they can maintain independence in daily activities. All participants must have scores above the threshold on cognitive screening tests like the ACE III and IFS, ensuring no significant cognitive impairment at the baseline.

The study will measure the effects of 5-MeO-DMT through a range of cognitive and psychiatric assessments:

Cognitive Assessments: These include the Rey Auditory Verbal Learning Test (RAVLT) for episodic memory, the Trail Making Test (TMT) for attention and cognitive flexibility, the Semantic and Phonological Fluency Test (SFT-FAS) for verbal fluency, the Paced Auditory Serial Addition Test (PASAT) for processing speed, and the Digit Span Subtests (DSS) for attention and working memory. These tests will provide valuable insights into how 5-MeO-DMT affects cognitive functions.

Psychiatric Assessments: These will assess symptoms of suicidal ideation (SSI), mood (BDI II), anxiety (STAI), and mindfulness (FFMQ), as well as self-reported cognitive complaints (CQC). These evaluations will help determine the psychological and emotional impact of 5-MeO-DMT on participants.

In addition, the study will include biochemical assessments such as microalbuminuria, blood glucose levels, liver and kidney function, cholesterol, and several biomarkers of inflammation. Cardiovascular evaluations will also be conducted during the trial, ensuring comprehensive monitoring of potential side effects.

This structured approach will help researchers assess the cognitive and psychological effects of 5-MeO-DMT in individuals with mild to moderate Alzheimer's disease. By focusing on participants with elevated anxiety, depression, and early cognitive decline, this trial aims to provide insights into the therapeutic potential of 5-MeO-DMT for neurodegenerative conditions.

DETAILED DESCRIPTION:
This Phase I/II clinical trial is designed to rigorously evaluate the efficacy of a novel sublingual formulation of 5-MeO-DMT in reducing symptoms of anxiety, depression, and cognitive decline in individuals diagnosed with mild to moderate Alzheimer's disease. The trial will employ a randomized, double-blind, placebo-controlled design, considered the gold standard in clinical research, to ensure unbiased and reliable results. By blinding both participants and investigators to treatment allocations, the study aims to generate robust data on the therapeutic potential of 5-MeO-DMT in this specific patient population.

Participants will be randomly assigned to one the placebo group or to the groups receiving 6 mg 5-MeO-DMT. Each dose group will include 10 participants, with a total of 20 volunteers enrolled. The dosing regimen consists of one sublingual administration per week over four consecutive weeks, allowing the study to assess both immediate and cumulative effects of 5-MeO-DMT on cognitive, mood, and anxiety symptoms.

Outcome Measures and Assessments: The primary outcome measure will focus on evaluating changes in cognitive function, mood, and anxiety symptoms, using a comprehensive set of neuropsychological and psychiatric assessments at multiple time points throughout the trial. Key cognitive assessments will include the Clinical Dementia Rating (CDR), Activities of Daily Living Questionnaire (ADLQ), and the Addenbrooke's Cognitive Examination III (ACE-III). These scales will provide a detailed overview of cognitive decline and the ability of 5-MeO-DMT to potentially mitigate these effects. Additionally, the Ineco Frontal Screening (IFS) will be administered to assess frontal lobe functioning.

Key psychiatric assessments will include the State-Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI), and Suicidal Ideation Scale (SSI), which are validated tools for measuring anxiety, depression, and suicidal thoughts. These assessments will help evaluate the emotional and psychological impact of 5-MeO-DMT on participants with Alzheimer's-related cognitive impairment.

Neurocognitive Assessments: To further evaluate the impact of 5-MeO-DMT on cognitive function, a battery of neurocognitive tests will be conducted. These will include the Rey Auditory Verbal Learning Test (RAVLT) to assess episodic memory, the Trail Making Test (TMT) for attention and cognitive flexibility, and the Digit Span Subtests (DSS) to measure working memory and attention. These tests will be administered at baseline, during dosing, and at the conclusion of the study (week 5) to monitor changes in cognitive function across time.

Study Design and Safety Measures: Safety will be closely monitored throughout the study. Regular assessments will be conducted to track vital signs, including heart rate, blood pressure, and temperature. Electrocardiograms (ECGs) will be taken to monitor any potential cardiovascular effects. Biochemical markers will be measured to assess any systemic effects, and psychological evaluations will be conducted to identify any changes in emotional or cognitive states that may signal adverse reactions or therapeutic benefits of the drug.

The findings from this study will offer valuable insights into the potential efficacy of sublingual 5-MeO-DMT in improving cognitive function and reducing symptoms of anxiety and depression in individuals with mild to moderate Alzheimer's disease. By focusing on participants with cognitive impairment and comorbid emotional symptoms, this trial aims to determine whether 5-MeO-DMT could be a beneficial treatment option for individuals suffering from both neurodegeneration and mental health disorders. The results will contribute to the growing body of evidence supporting the use of psychedelic compounds in treating cognitive decline, anxiety, and depression, providing new possibilities for managing Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 80 years
* Diagnosis of mild to moderate Alzheimer's disease
* Clinical Dementia Rating (CDR) score between 0.5 and 1
* ACE-III score ≤ 86 for individuals with high educational levels (≥12 years of schooling)
* ACE-III score < 62 for individuals with low educational levels (≤12 years of schooling)
* Moderate to high levels of anxiety, as defined by:
* State-Trait Anxiety Inventory (STAI-S) State score ≥20 for men, ≥23 for women
* STAI-Trait score ≥20 for men, ≥26 for women
* Mild to moderate depressive symptoms, as indicated by a Beck Depression Inventory (BDI) score ≥21
* Must provide written informed consent to participate in the study

Exclusion Criteria:

* Liver dysfunction
* Cardiovascular conditions (e.g., uncontrolled hypertension, angina, significant ECG abnormalities, recent transient ischemic attack or stroke, peripheral/pulmonary vascular disease without active claudication).
* Blood pressure >140 mmHg systolic or >90 mmHg diastolic
* Epilepsy or history of seizures
* Kidney failure
* Insulin-dependent diabetes
* Chronic obstructive pulmonary disease (COPD)
* Increased intracranial or cerebrospinal pressure
* Hyperthyroidism
* Psychotic symptoms or family history of psychotic disorders
* Prodromal symptoms of schizophrenia or dissociative identity disorder
* Severe depression or anxiety requiring immediate treatment with antidepressants or daily anxiolytics, particularly in cases with suicidal ideation
* Medications: Regular use of psychoactive medications, including benzodiazepines, serotonin-active medications (e.g., ondansetron), or monoamine oxidase inhibitors (MAOIs)
* Drug Interactions: Use of potent metabolic inducers or inhibitors, such as: Inducers: rifampicin, anticonvulsants (e.g., carbamazepine, phenytoin), nevirapine, efavirenz, taxol, dexamethasone. Inhibitors: HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, troleandomycin.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Phonological Verbal Fluency Test (FAS) from Baseline to Week 5 | The FAS will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess changes in executive function during and after sublingual 5-MeO-DMT administration.
  The Phonological Verbal Fluency Test (FAS) measures executive function by assessing a participant's ability to generate words within a specific time limit, categorized by a starting letter. The task is designed to evaluate verbal memory, cognitive flexibility, and processing speed. A higher score indicates better performance.
Change in Paced Auditory Serial Addition Test (PASAT) from Baseline to Week 5 | The PASAT will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to evaluate the effects of 5-MeO-DMT on cognitive processing speed and attention.
  The Paced Auditory Serial Addition Test (PASAT) is a cognitive test used to measure processing speed and attention. Participants are presented with a sequence of numbers and must add each new number to the previous one as quickly as possible. Performance is scored based on the number of correct responses within a given time. A higher score reflects better cognitive processing and attention.
Change in Digit Span Scale (DSS) from Baseline to Week 5 | The DSS will be administered at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess changes in attention and working memory following 5-MeO-DMT administration.
  The Digit Span Scale (DSS) is used to assess attention span and working memory. In this test, participants must repeat a series of numbers either in the same order (forward) or in reverse (backward). The DSS measures short-term memory and cognitive flexibility. A higher score indicates better working memory and attention capacity.
Mystical Experience Questionnaire (MEQ) Assessment at 40 Minutes Post-Administration | The MEQ will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to assess the subjective mystical experiences induced by sublingual 5-MeO-DMT.
  The Mystical Experience Questionnaire (MEQ) is used to assess the subjective mystical experiences following psychedelic administration. It evaluates aspects such as feelings of unity, transcendence, and the sense of the sacred. The MEQ includes questions about altered perceptions of time, space, and self, as well as emotional and cognitive shifts. Higher scores indicate a stronger experience of mystical qualities.
Peak Experience Scale (PES) Assessment at 40 Minutes Post-Administration | The PES will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to capture the intensity and emotional impact of the 5-MeO-DMT experience.
  The Peak Experience Scale (PES) is a tool for measuring the intensity and quality of peak experiences following psychedelic use. It includes items related to emotional intensity, personal insight, and transcendence. Participants rate the emotional and psychological impact of their experiences, with higher scores reflecting more intense peak experiences.
Ego Dissolution Inventory (EDI) Assessment at 40 Minutes Post-Administration | The EDI will be completed at 40 minutes post-administration during each dosing week (Weeks 1-4) to evaluate the degree of ego dissolution experienced after 5-MeO-DMT consumption.
  The Ego Dissolution Inventory (EDI) assesses the extent to which participants experience a loss of ego boundaries or self-identity following psychedelic administration. It includes questions that explore the feeling of oneness with the environment, other people, or the universe, as well as the dissolution of self-related thoughts and ego. Higher scores indicate stronger experiences of ego dissolution.

SECONDARY OUTCOMES:
Mean change in Beck Depression Inventory II (BDI-II) from Baseline to Week 5 | The BDI-II will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess the impact of 5-MeO-DMT on the severity of depression.
  The Beck Depression Inventory II (BDI-II) is a 21-item self-report questionnaire designed to assess the severity of depressive symptoms. Each item is scored from 0 to 3, with the total score ranging from 0 to 63. Higher scores indicate more severe depression.
Mean change in State-Trait Anxiety Inventory (STAI) from Baseline to Week 5 | STAI evaluations will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to assess the impact of 5-MeO-DMT on anxiety levels.
  The State-Trait Anxiety Inventory (STAI) is a 40-item scale that measures both state anxiety (current feelings of anxiety) and trait anxiety (general tendency to experience anxiety). Each item is scored from 1 to 4, with the overall score ranging from 20 to 80. Higher scores indicate higher levels of anxiety.
Mean change in Depression, Anxiety, and Stress Scale (DASS-21) from Baseline to Week 5 | DASS-21 will be conducted at baseline (Week 0), during treatment (Weeks 1-4), and at follow-up (Week 5) to evaluate the impact of 5-MeO-DMT on mood and stress.
  The Depression, Anxiety, and Stress Scale (DASS-21) is a 21-item questionnaire that measures the severity of depression, anxiety, and stress symptoms. Each item is scored from 0 to 3, with higher scores indicating more severe symptoms. The total score ranges from 0 to 63.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Bruno, PhD, Study Chair — Biomind Labs Inc.
Locations (1):
- Hospital Descentralizado Dr. Marcial V. Quiroga., San Juan, Rivadavia, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The study is committed to advancing scientific research by planning to share individual participant data (IPD) to contribute valuable insights to the research community. We will provide a detailed data dictionary alongside the IPD, outlining the variables and types of data collected for each participant, facilitating comprehensive analysis by researchers.
  Specifically, we plan to share all IPD collected throughout the trial, including data that underlie published results. Importantly, all personal information and identifying details of participants will remain strictly confidential and will not be disclosed. This commitment ensures the privacy of individuals involved while enabling meaningful contributions to scientific knowledge.
Supporting Information: Study Protocol, ICF
Time Frame: The individual participant data (IPD) and any supporting information will be made available starting 6 months after the publication of the study results. This will allow sufficient time for data analysis and the dissemination of primary findings. The data will remain available for at least 5 years following the publication, ensuring ample time for other researchers to access and utilize the data for further analysis or related studies. In case of any modifications to the availability period, these will be communicated clearly along with the reasons. This time frame is subject to ethical and regulatory requirements and may be adjusted if necessary.
Access Criteria: Researchers seeking access to the individual participant data (IPD) and supporting information must submit a formal request outlining their proposed analyses. This proposal should detail the types of analyses, including the statistical methods to be used, which will be reviewed for scientific merit and methodological rigor. A signed data sharing agreement will be required, and the request must be submitted through the designated data sharing platform or by email to the study's data management team. Access to IPD will be granted based on ethical review and approval, ensuring that the proposed research aligns with the study's objectives and respects participant confidentiality. All requests will be reviewed by an independent committee responsible for overseeing data sharing, ensuring transparency, and safeguarding participant privacy.

REFERENCES:
- See also: Biomind Labs is developing the next generation of pharmaceuticals to treat patients suffering from neurological disorders. This unique approach targets the original and initial drivers of the diseases. — https://www.biomindlabs.com/